CLINICAL TRIAL: NCT01194323
Title: Biology in Patients With Reflux Esophagitis and Mucosal Impedance
Brief Title: Biology in Patients With Reflux Esophagitis
Acronym: BENCH
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Medical Director, Vanderbilt University Medical Center
Other Study IDs: BENCH
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: GERD
Keywords: esophageal erosion; abnormal pH monitoring
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total RNA and proteins will be extracted from de-identified samples. Genes' and proteins' expression will be processed and analyzed at Vanderbilt Core Facilities.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: No complaints or history of heartburn or acid regurgitation; no erosion at EGD; and normal pH monitoring
- GERD Cases: Patients with esophageal erosion at EGD and abnormal pH monitoring.

SUMMARY:
GERD is a common condition in the western world. In most cases, the diagnostic is established by good response to empiric proton pump inhibitor (PPI) therapy. When the patient symptoms are refractory to therapy, multiple invasive tests are available. The results of those tests (EGD, manometry, Ph monitoring and impedance) are clues that the physician use together to establish the diagnostic. No test however can be use alone because of their poor specificity and sensitivity. Recently, microscopy has been used to detect dilated intercellular space in between distal esophageal cells tissue; unfortunately this marker again failed to diagnose GERD.

In search of more sensitive and specific markers of GERD, we propose to assess if acid exposure affects: 1) gene and proteins expression in the esophageal/post-cricoid area tissue; and 2) local impedance of the mucosa. The secondary aim of this proposal is to determine if correlation exists between the two approaches.

ELIGIBILITY:
Inclusion Criteria (GERD Cases):

* Male or female
* Ages 18 years or older
* Undergoing EGD as standard of care at Vanderbilt's Digestive Diseases Center
* Esophageal erosion detected at EGD
* Abnormal pH monitoring

Inclusion Criteria (Controls):

* Male or female
* Ages 18 years or older
* Undergoing EGD as standard of care at Vanderbilt's Digestive Diseases Center
* No complaints or history o heartburn or acid regurgitation
* No erosion at EGD
* Normal pH monitoring

Exclusion Criteria:

* Less than 18 years of age
* Unable to provide informed consent
* Use of acid suppressive therapy within last 14 days
* known history of Barrett's esophagus, gastric surgery, alcoholism, significant motility condition
* contraindications to biopsy such as taking anticoagulants other than aspirin (coumadin, plavix) or allergies to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female volunteers ages 18 years and older; able to give informed consent; no use of acid suppressive therapy within 14 days prior to procedure; no history of Barret's esophagus, gastric surgery, alcoholism, or significant motility condition; no contraindications to biopsy, including taking anticoagulants or allergies to local anesthetic.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in gene and protein expression due to acid exposure in the esophagus | Chronic exposure
  We are assessing if acid exposure affects gene and protein expression in the esophageal/post-cricoid area tissue
Change in local impedance of the esophageal mucosa | Chronic exposure
  We are assessing if acid exposure affects local impedance of the mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaezi, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Digestive Diseases Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saritas Yuksel E, Higginbotham T, Slaughter JC, Mabary J, Kavitt RT, Garrett CG, Vaezi MF. Use of direct, endoscopic-guided measurements of mucosal impedance in diagnosis of gastroesophageal reflux disease. Clin Gastroenterol Hepatol. 2012 Oct;10(10):1110-6. doi: 10.1016/j.cgh.2012.05.018. Epub 2012 May 27. PMID 22642956